CLINICAL TRIAL: NCT03962933
Title: Urine-based Detection of Non-muscle Invasive Bladder Cancer Recurrence
Brief Title: Urine-based Detection of Non-muscle Invasive Bladder
Acronym: SOLUSION
Status: Completed | Type: Observational
Sponsor: Nessn Azawi (Other)
Responsible Party: Sponsor-Investigator, Nessn Azawi, Associate professor, Zealand University Hospital
Organization: Zealand University Hospital (Other)
Other Study IDs: SOLUSION
Record Dates: First submitted 2019-05-23; First posted 2019-05-24 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Flexcystoscopy/Uromonitor: Control cystoscopy every 4 - 8 and 12 months as a standard procedure, And Urine test (Uromonitor) every 4 months

SUMMARY:
Non-muscle invasive bladder cancer (NMIBC), which comprises approximately 75% of bladder tumors, has the highest recurrence rate of all cancers, with around 70% of the patients developing local recurrences, despite elaborated treatments. Uromonitor is a completely Non-Invasive urine based IVD diagnosis test. It´s able to detect Non-muscle invasive bladder cancer with 100% sensitivity and 97,3 % specificity. Regardless of Tumor stage and grade (unlike Cytology). The rate of Uromonitor false positives (2,3%) is actually lower than the rate of Cystoscopy false positives (3,5%).

DETAILED DESCRIPTION:
Non-muscle invasive bladder cancer (NMIBC), which comprises approximately 75% of bladder tumors, has the highest recurrence rate of all cancers, with around 70% of the patients developing local recurrences, despite elaborated treatments. Uromonitor is a completely Non-Invasive urine based IVD diagnosis test. It´s able to detect Non-muscle invasive bladder cancer with 100% sensitivity and 97,3 % specificity. Regardless of Tumor stage and grade (unlike Cytology). The rate of Uromonitor false positives (2,3%) is actually lower than the rate of Cystoscopy false positives (3,5%).

Hypothesis:

The study aims at evaluating the potential clinical impact of a highly sensitive urinary marker, Uromonitor, regarding possible reduction in number of cystoscopies.

We hypothesize that the use of a sensitive urinary marker regarding recurrent tumor will enable us to reduce the number of follow-up cystoscopies without risk of delaying diagnosis of recurrence and progression cystoscopies compared to flexible cystoscopy alone.

We hypothesize that number of tumors missed at follow-up cystoscopy alone or urinary marker alone is identical or in favor of a sensitive urinary marker that can detect sub-visible lesions and the examinations combined identify all tumor recurrences.

Moreover, we hypothesize that tumors missed at follow-up at a given time point are very small and will be identified at next follow-up without increasing the risk of progression and that regular follow-up with cystoscopy alone therefore can be replaced by follow-up with a sensitive urinary biomarker alone - where cystoscopy only is performed if the biomarker is positive.

ELIGIBILITY:
Inclusion Criteria:

* Patients who previously had low grad NMIBC.
* Subjects must provide written informed consent prior to performance of study-specific procedures or assessments, and must be willing to comply with treatment and follow-up.

Exclusion Criteria:

* Clinical suspicion of muscle invasive bladder cancer
* Upper urinary track tumours
* Patients undergoing neoadjuvant chemotherapy based on local protocols
* Metastatic urothelial carcinoma
* Patients recived installation therapy within the last 4 weeks

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: on-muscle invasive bladder cancer (NMIBC), which comprises approximately 75% of bladder tumors, has the highest recurrence rate of all cancers, with around 70% of the patients developing local recurrences, despite elaborated treatments. Uromonitor is a completely Non-Invasive urine based IVD diagnosis test. It´s able to detect Non-muscle invasive bladder cancer with 100% sensitivity and 97,3 % specificity. Regardless of Tumor stage and grade (unlike Cytology). The rate of Uromonitor false positives (2,3%) is actually lower than the rate of Cystoscopy false positives (3,5%).
Sampling Method: Probability Sample
Enrollment: 196 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Recurrences rate | 5 years
  Recurrences rate

CONTACTS AND LOCATIONS:
Locations (1):
- Zealand University Hospital, Roskilde, Denmark

IPD SHARING:
Plan to Share IPD: No